CLINICAL TRIAL: NCT02990741
Title: A Randomized Clinical Trial on Atrial Fibrillation Screening by Using an Automated Electrocardiogram System in an Elderly Chinese Population
Brief Title: A Clinical Trial Screening for Atrial Fibrillation (AF-CATCH)
Acronym: AF-CATCH
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Shanghai Jiao Tong University School of Medicine
Other Study IDs: AF-CATCH
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; automated ECG system
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Usual screening group: ECG recordings at baseline plus at 1 and 2 year of follow-up; three ECG recordings in total.
- Intensive screening subgroup: ECG recordings at baseline plus quarterly during follow-up, at months 3, 6, 9 ,12, 15, 18, 21 and 24; 9 ECG recordings in total.
- More intensive screening subgroup: ECG recordings at baseline plus weekly during the first month of follow-up and quarterly afterwards, at weeks 1, 2, 3 and 4 and months 3, 6, 9, 12, 15, 18, 21 and 24; 13 ECG recordings in total.

SUMMARY:
1. Study name:A randomized clinical trial on atrial fibrillation screening by using an automated electrocardiogram system in an elderly Chinese population
2. Rationale: Failure in the diagnosis and management of atrial fibrillation leads to high incidence of stroke and high mortality and disability. It is therefore imperative to diagnose and manage atrial fibrillation in a timely and effective fashion to prevent the complications of atrial fibrillation.
3. Objective:The primary objective is to investigate whether more frequent ECG recordings and analyses with this automated ECG system (4 times/year) would significantly improve the detection of atrial fibrillation compared to a single annual ECG screen.The secondary objective is to explore whether even more frequent ECG recordings and analyses (8 times/year) would further improve the detection of atrial fibrillation.
4. Study design: The present study is designed as a randomized controlled trial of parallel group (two).
5. Study population: Men and women aged at least 65 years (n=7000) meet the inclusion/exclusion criteria.
6. Randomization and treatment: Eligible subjects will be randomized in a 1:1 ratio into the usual and intensive screening groups with 3500 patients in each group, and within the intensive screening group in a 3:1 ratio into the intensive and more intensive subgroups with 2625 and 875 patients, respectively.
7. Follow up: 1)Usual screening group: ECG recordings at baseline plus at 1 and 2 year of follow-up; three ECG recordings in total. 2)Intensive screening subgroup: ECG recordings at baseline plus quarterly during follow-up, at months 3, 6, 9, 12, 15, 18, 21 and 24; 9 ECG recordings in total. 3)More intensive screening subgroup: ECG recordings at baseline plus weekly during the first month of follow-up and quarterly afterwards, at weeks 1, 2, 3 and 4 and months 3, 6, 9, 12, 15, 18, 21 and 24; 13 ECG recordings in total.
8. Sample size estimation: The number of required subject for the whole trial is 7000.
9. Timeline: Start of subjects enrollment : December 2016; End of subjects enrollment : June 2017; End of study : October 2020
10. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

DETAILED DESCRIPTION:
1. Study name:A randomized clinical trial on atrial fibrillation screening by using an automated electrocardiogram system in an elderly Chinese population
2. Rationale: The incidence of atrial fibrillation rises continuously.The main detrimental effect of atrial fibrillation is its complication of stroke.Failure in the diagnosis and management of atrial fibrillation before the incidence of stroke leads to high mortality and disability. It is therefore imperative to diagnose and manage atrial fibrillation in a timely and effective fashion and prevent the complications of atrial fibrillation, by screening followed by the use of proven therapy, such as warfarin. An automated handheld ECG system based on a smartphone has recently become available for the screening of atrial fibrillation in high risk people.However, how this system can be most effectively used for the widespread screening of atrial fibrillation remains a question that requires investigation. Moreover, while repeated recordings will have a higher yield of atrial fibrillation diagnosis [11], it is not certain what constitutes an optimum number of ECG recordings balancing cost and effectiveness. The present study was therefore designed as a randomized controlled trial to investigate whether more frequent ECG recordings and analyses with this automated ECG system would significantly improve the detection of atrial fibrillation compared to a single annual ECG screen in elderly Chinese population in the community health centre.
3. Objective:The primary objective is to investigate whether more frequent ECG recordings and analyses with this automated ECG system (4 times/year) would significantly improve the detection of atrial fibrillation compared to a single annual ECG screen.The secondary objective is to explore whether even more frequent ECG recordings and analyses (8 times/year) would further improve the detection of atrial fibrillation.
4. Study design: The present study is designed as a randomized controlled trial of parallel group (two)
5. Study population: Men and women aged at least 65 years (n=7000) will be recruited from 5 community health centers in the city of Shanghai. Eligible patients should meet the following inclusion and exclusion criteria.Inclusion Criteria:1) Age≥65 years; 2) Absence of atrial fibrillation at baseline; 3) Willing and capable to visit the outpatient clinic on his/her own for long-term follow-up. Exclusion Criteria:1) Known persistent or paroxysmal atrial fibrillation : Sinus rhythm after pharmacological or electric cardioversion, or radiofrequency ablation;Use of anticoagulant therapy and atrial fibrillation;Use of medication for heart rate control;Untreated atrial fibrillation.2) Serious life-threatening diseases, such as, cancer, severe cardiac, cerebral, liver, kidney diseases, etc;3) Difficult for long-term follow-up visit for any reason
6. Randomization and treatment: Eligible subjects will be randomized in a 1:1 ratio into the usual and intensive screening groups with 3500 patients in each group, and within the intensive screening group in a 3:1 ratio into the intensive and more intensive subgroups with 2625 and 875 patients, respectively. 1)Usual screening group: ECG recordings at baseline plus at 1 and 2 year of follow-up; three ECG recordings in total. 2)Intensive screening subgroup: ECG recordings at baseline plus quarterly during follow-up, at months 3, 6, 9,12, 15, 18, 21 and 24; 9 ECG recordings in total. 3)More intensive screening subgroup: ECG recordings at baseline plus weekly during the first month of follow-up and quarterly afterwards, at weeks 1, 2, 3 and 4 and months 3, 6, 9, 12, 15, 18, 21 and 24; 13 ECG recordings in total. The automated electrocardiogram analysis system AliveCor® Heart Monitor will be used to perform ECG recordings and analysis for the immediate diagnosis of atrial fibrillation. At one and two year of follow-up, a follow-up questionnaire will be administered and physical examinations will be performed. All detected cases of atrial fibrillation will be further evaluated with a regular 12-lead ECG, and then referred to a specialists' centre for treatment.
7. Follow up: In the usual screening group, patients will be followed-up in the community health centre at baseline and at 12 and 24 months of follow-up. In the intensive screening group, patients will be followed-up at baseline and at 3, 6, 9, 12, 15, 18, 21 and 24 months of follow-up. In the more intensive screening subgroup, patients will be followed-up weekly in the first month of follow-up and at 3, 6, 9, 12, 15, 18, 21 and 24 months of follow-up.
8. Sample size estimation: The detection rate of atrial fibrillation by a single 12-lead ECG was 2.5% in elderly people living in Shanghai Of the 2.5%, only 0.5% were aware of atrial fibrillation. The detection rate of atrial fibrillation by an ECG recording at baseline and another in 12 months could be estimated to be 2.0% in elderly people without awareness of atrial fibrillation. The primary hypothesis is that the detection rate could be improved by 50% with more frequent ECG recordings. If =0.05, power=80% and one-sided test are assumed, and a 1:1 ratio would be used to assign patients to usual and intensive ECG screening, the study will require a sample size of 3013 subjects per group. In consideration of a 15% of super-addition, approximately 3500 eligible subjects per group should be enrolled. The number of required subjects for the whole trial is 7000.
9. Timeline : Enrollment rate : 1000 patients /month ; Planned publication /presentation : October 2020; Start of subjects enrollment : December 2016; End of subjects enrollment : June 2017; End of study : October 2020
10. Organization: The study will be conducted in a single research center (Ruijin Hospital) with 5 community health centers. Patients will be recruited and followed up by the community health physicians in 5 community health centers, under the supervision of cardiologists from Ruijin Hospital. ECG will be recorded in each of the community health centers. Atrial fibrillation will be initially diagnosed by the software build in the smart phone. ECG will also be transmitted to a cloud platform for storage and further analysis. If atrial fibrillation is detected, a 12-lead ECG will be immediately performed for the verification and confirmation of the diagnosis of atrial fibrillation. The identified patients with atrial fibrillation will be referred to the outpatient clinic of Ruijin Hospital for management.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years;
2. Absence of atrial fibrillation at baseline;
3. Willing and capable to visit the outpatient clinic on his/her own for long-term follow-up.

Exclusion Criteria:

1. Known persistent or paroxysmal atrial fibrillation 1)Sinus rhythm after pharmacological or electric cardioversion, or radiofrequency ablation; 2)Use of anticoagulant therapy and atrial fibrillation; 3)Use of medication for heart rate control; 4)Untreated atrial fibrillation.
2. Serious life-threatening diseases, such as, cancer, severe cardiac, cerebral, liver, kidney diseases, etc;
3. Difficult for long-term follow-up visit for any reason.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men and women aged at least 65 years (n=7000) will be recruited from 5 community health centers in the city of Shanghai and randomized into a group of more frequent (4 or 8) ECG recordings and analyses (n=3500) and a group of a single ECG recording and analysis during 12 months of follow-up (n=3500). The intensive screening group will be further randomly divided into intensive (n=2625) and more intensive subgroups (n=875). Eligible patients should meet the following inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 4348 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Difference in the detection rate of atrial fibrillation between the usual and the intensive screening groups | 2 year

SECONDARY OUTCOMES:
Difference in the detection rate of atrial fibrillation between the intensive and more intensive screening subgroups within the intensive group | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, MD, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang W, Chen Y, Miao CY, Huang QF, Sheng CS, Shao S, Wang D, Xu SK, Lei L, Zhang D, Chen YL, Hu LX, Xia JH, Ye XF, Cheng YB, Wang Y, Guo QH, Li Y, Lowres N, Freedman B, Wang JG; AF-CATCH Investigators and Coordinators. Quarterly versus annual ECG screening for atrial fibrillation in older Chinese individuals (AF-CATCH): a prospective, randomised controlled trial. Lancet Healthy Longev. 2021 Aug;2(8):e470-e478. doi: 10.1016/S2666-7568(21)00138-0. Epub 2021 Jul 23. PMID 36097996
- [Derived] Zhang W, Chen Y, Hu LX, Xia JH, Ye XF, Cheng YB, Wang Y, Guo QH, Li Y, Lowres N, Freedman B, Wang JG; AF-CATCH Investigators and Coordinators. Changes in the CHA2DS2-VASC score as a predictor of incident atrial fibrillation in older Chinese individuals: the AF-CATCH study. Eur Heart J Open. 2022 Jul 25;2(4):oeac046. doi: 10.1093/ehjopen/oeac046. eCollection 2022 Jul. PMID 35983405